CLINICAL TRIAL: NCT05957107
Title: Randomized, Double-blind, Placebo, Positive-controlled Phase II Trial of VDJ001 in Patients With Moderate-to-severe Active Rheumatoid Arthritis
Brief Title: Phase II Trial of VDJ001 in Patients With Moderate-to-severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing VDJBio Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VDJ001-RA-II
Record Dates: First submitted 2023-07-11; First posted 2023-07-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Injection of recombinant humanized monoclonal antibody against interleukin-6 receptor 4 mg/kg (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 4 mg/kg as the low dose group.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection
- Injection of recombinant humanized monoclonal antibody against interleukin-6 receptor6mg/kg (Experimental): Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection 6mg/kg as the middle dose group.
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection
- placebo control (Experimental): placebo control
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection
- Tocilizumab Injection8mg/kg (Experimental): Tocilizumab Injection8mg/kg
  Interventions: Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection

INTERVENTIONS:
Biological: Recombinant Humanized Anti-interleukin-6 Receptor Monoclonal Antibody Injection — The drug was administered once every 4 weeks.
  Other Names: Tocilizumab Injection; placebo control

SUMMARY:
This is a multicenter, randomized, double-blind, placebo and tocilizumab controlled phase II trial in RA patients to evaluate the initial efficacy, safety, pharmacokinetic, pharmacodynamic characteristics, and immunogenicity of VDJ001 in RA patients.

DETAILED DESCRIPTION:
After screening, eligible subjects were randomly assigned in a 1:1:1:1 ratio to VDJ001 4 mg/kg group, VDJ001 6 mg/kg group, placebo group, and tocilizumab group to receive trial drug or control drug every 4 weeks. The treatment course was 12 weeks (D1, W4, W8 administration, followed up to W12).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be included:

  1. Voluntarily sign the informed consent;
  2. Age 18-75 years old (including boundary values);
  3. RA was diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 ACR and EULAR classification criteria;
  4. Moderate to severe active RA was determined according to the following criteria: the number of joint swelling ≥6 (based on 66 joints) and the number of joint tenderness ≥6 (based on 68 joints), and the C-reactive protein (CRP) ≥10 mg/L or erythrocyte sedimentation rate (ESR) ≥28 mm/h;
  5. Had received oral methotrexate (MTX) therapy for at least 12 weeks with a stable dose (MTX dose of 7.5-25 mg/ week) for at least 4 weeks before randomization; Subjects with a history of parenteral MTX use (subcutaneous, intramuscular, or intravenous) were eligible, but they had to have received a stable dose of MTX 7.5 to 25mg/ week orally for ≥4 weeks before randomization;
  6. If subjects were taking prednisone or equivalent glucocorticoids at the time of screening, they were treated with a stable dose (prednisone dose ≤10mg/ day) for at least 4 weeks before randomization.

     Exclusion Criteria:

     Participants who meet any of the following conditions will not be included in the study:

  <!-- -->

  1. Weight >100 kg or <40 kg.
  2. Patients with ACR function grade IV or long-term bedridden/wheelchair-bound.
  3. Persons with allergies or known allergies to any of the ingredients and/or other similar products under study.
  4. The investigator determined that the subject had undergone or planned surgery that might affect the study evaluation of the evaluated joint.
  5. Patients with rheumatic immune diseases other than rheumatoid arthritis, uncontrolled immune system diseases requiring oral corticosteroid treatment, were considered by the investigators to influence trial evaluators.
  6. Primary or secondary immunodeficiency (previous or current active).
  7. Previous or current cancer.
  8. A history of any lymphoproliferative disease, such as EBV-associated lymphoproliferative disease, lymphoma, leukemia, myeloproliferative disease, multiple myeloma, or signs and symptoms suggestive of current lymphoproliferative disease.
  9. The presence of serious, poorly controlled concomitant diseases, such as (but not limited to) neurological, cardiovascular, hepatic, renal, gastrointestinal, and endocrine diseases, which in the judgment of the investigator may prevent the subjects from participating in the study.
  10. Have any congenital or acquired neurological disease, vascular disease, or systemic disease, especially joint pain and swelling (e.g., Parkinson's disease, cerebral palsy, diabetic neuropathy) that may affect the evaluation of the effectiveness of this study.
  11. The following infections are known: Recurrent active bacteria, viruses, fungi, mycobacteria infection or other (including but not limited to, and atypical mycobacteria tuberculosis disease, chest X-ray examination showed granulomatous disease, hepatitis c virus (HCV) infection, HIV infection, herpes zoster, but does not include the nail bed fungus infection), or 6 months before the filter has a history of chronic infection, Or any major episode of infection requiring hospitalization or intravenous antibiotic treatment within 4 weeks prior to screening or oral antibiotic treatment within 2 weeks prior to screening, or a history of tuberculosis; For those who screened positive for TB, enrollment was determined by the investigator after prophylactic treatment.
  12. Subjects who received live/attenuated/inactivated COVID-19 vaccine within 4 weeks prior to the screening visit or were known to receive live/attenuated/inactivated COVID-19 vaccine during the 12-week treatment observation period.
  13. Patients who had used lymphocyte depletion agents/therapies, alkylating agents, total lymphoid irradiation, or other therapies before screening or planned to use them during the study.
  14. Previous treatment with IL-6 and IL-6R inhibitors.
  15. Use biological DMARDs at the following times:

      A) Anapheresis, etanercept: within 28 days before administration;

      B) Adalimumab, infliximab: within 56 days before administration;

      C) Golimumab and cetuzumab: within 70 days before administration;

      D) Abacept: within 84 days before administration;

      E) Denoxemide: within 150 days before administration;

      F) Rituximab: within 180 days before administration.
  16. Abiotic DMARDs other than MTX were administered within 28 days prior to dosing (subjects without chloroquine, hydroxychloroquine, leflunomide within 56 days prior to dosing, or no more than 28 days after standard koleenamine treatment or active carbon washout were not eligible).
  17. Had received intra-articular or extra-intestinal corticosteroid therapy within 28 days prior to dosing.
  18. Who had been immunized with genofin, gold thiodextrose (gold for injection), gold thiomalate (gold for injection), or oral polio vaccine within 56 days prior to administration.
  19. Patients who received intravenous immunoglobulin, plasma exchange or Prosorba column within 24 weeks before screening.
  20. Participated in clinical studies of other drugs within 1 month prior to screening or within 5 half-lives of other experimental drugs, whichever is longer.
  21. Hepatitis B surface antigen (HBsAg) positive, or if hepatitis B core antibody (HBcAb) positive, HBV DNA test is added and HBV DNA> the lower limit of detection.
  22. The laboratory test value (retest is allowed, and the last test result shall prevail) meets any of the following conditions:

      • Serum creatinine: female subjects had serum creatinine >1.4 mg per deciliter (124 μmol per liter); Serum creatinine > 1.6 mg/dL (141 μmol/L) in male subjects;

      ALT or AST> 1.5 times the upper limit of normal (ULN);
      * Platelet count <80×109/ L;
      * the WBC < 3.5 x 109 / L;
      * Total bilirubin > 1.5 times ULN.
  23. Female subjects who had a positive pregnancy test during pregnancy, or breastfeeding, or screening, or who were unable to use effective contraception from the screening period until 6 months after completion or termination of the trial (including male subjects and their female spouses).
  24. Other ineligible subjects were judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieved ACR20 at week 12. | 12 weeks
  Proportion of patients who achieved American College of Rheumatology 20% improvement criteria (ACR20) at week 12.

SECONDARY OUTCOMES:
Proportion of patients who achieved ACR50, ACR70 at week 12. | 12 weeks
  Proportion of patients who achieved American College of Rheumatology 50%, 70% improvement criteria at week 12.
Proportion of patients who achieved DAS28-CRP <2.6, DAS28-ESR <2.6, DAS28-CRP <3.2, DAS28-ESR <3.2 at week 12. | 12 weeks
  DAS28-CRP=0.56*(TJC28)1/2+0.28*(SJC28)1/2+0.014*GH+0.36*ln(CRP+1)+0.96; DAS28-ESR=0.56*(TJC28)1/2+0.28*(SJC28)1/2+0.014*GH+0.70*ln(ESR); In the formula, TJC28 = joint count of pressure and pain at 28 joints, SJC28 = joint count of swelling at 28 joints, GH = general health status, i.e., patient's overall assessment of disease activity, ln = natural logarithm.
Proportion of patients who achieved a good response rate on the Clinical Disease Activity Index (CDAI) (defined as ≥50% improvement in CDAI or CDAI ≤2.8) at Week 12. | 12 weeks
  CDAI=TJC28+SJC28+PGA+PhGA In the formula, TJC28 = joint counts of pressure and pain at 28 joints, SJC28 = joint counts of swelling at 28 joints,PhGA stands for physician's global visual analogue scale of disease activity in cm, and PtGA stands for patient's global visual analogue scale of disease activity in cm.
Change in duration of morning stiffness at week 12 relative to baseline and rate of change. | 12 weeks
  Morning stiffness refers to the phenomenon that the diseased joints are stiff for a longer period of time in the morning after standing still, such as the feeling of glue, which is gradually reduced after appropriate activities.
Patient ratings of arthralgia | 12 weeks
  Change in patient rating of arthralgia (PtAAP) at week 12 relative to baseline and rate of change.
Patient's overall assessment of the condition | 12 weeks
  Patient's overall assessment of the condition (PtGA) at week 12 change from baseline and rate of change.
Physician's Global Assessment of Condition | 12 weeks
  Change in Physician's Global Assessment of Condition (PhGA) relative to Baseline and Rate of Change at Week 12.
Patient Health Assessment Questionnaire | 12 weeks
  Change in Patient Health Assessment Questionnaire (HAQ-DI) Score Relative to Baseline and Rate of Change at Week 12.
Health Status Questionnaire (SF-36) | 12 weeks
  Change from baseline in Week 12 Health Status Questionnaire (SF-36) scores and rate of change.
Functional Assessment of Chronic Illness Therapy-Fatigue Scale | 12 weeks
  Change from baseline and rate of change in Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) score at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Zhan-guo Li, Principal Investigator — Peking University People's Hospital
Locations (15):
- China (15):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Baoji Central Hospital, Baoji
  - Beijing Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Chenzhou First People's Hospital, Chenzhou
  - Pingxiang People's Hospital, Jiangxi
  - Jilin Province People's Hospital, Jilin
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing
  - Puyang Oilfield General Hospital, Pujiang
  - Qilu Hospital of Shandong University, Shandong
  - Peking University Shenzhen Hospital, Shenzhen
  - People's Hospital of Xinjiang Uygur Autonomous Region, Xinjiang
  - Zaozhuang Municipal Hospital, Zaozhuang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No